CLINICAL TRIAL: NCT06840691
Title: A Randomized, Open-lable, Single-dose, 3-sequence, 3-period Crossover Bioequivalence Study of Two Different PEG-rhGH （2mg/mL）Preparations in Chinese Healthy Adults
Brief Title: A Bioequivalence Study of Two Different Processes of PEG-rhGH Preparations
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GenSci034-102
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Growth Hormone Deficiency (PGHD)
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-R-R (Experimental): Administration order: PEG-rhGH with new preparation (T), PEG-rhGH with present preparation (R), PEG-rhGH with present preparation (R)
  Interventions: Drug: PEG-rhGH with new preparation (T); Drug: PEG-rhGH with present preparation (T)
- R-T-R (Experimental): Administration order: PEG-rhGH with present preparation (R), PEG-rhGH with new preparation (T), PEG-rhGH with present preparation (R)
  Interventions: Drug: PEG-rhGH with new preparation (T); Drug: PEG-rhGH with present preparation (T)
- R-R-T (Experimental): Administration order: PEG-rhGH with present preparation (R), PEG-rhGH with present preparation (R), PEG-rhGH with new preparation (T)
  Interventions: Drug: PEG-rhGH with new preparation (T); Drug: PEG-rhGH with present preparation (T)

INTERVENTIONS:
Drug: PEG-rhGH with new preparation (T) — A single subcutaneous injection of PEG-rhGH with new preparation
Drug: PEG-rhGH with present preparation (T) — A single subcutaneous injection of PEG-rhGH with present preparation

SUMMARY:
The purpose of this study is to investigate whether PEG-rhGH with new preparation is bioequivalent to PEG-rhGH with present preparation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether PEG-rhGH with new preparation is bioequivalent to PEG-rhGH with present preparation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged ≥18 years old and≤45 years old;
* The Body mass index (BMI): 19-26 kg/m2 (inclusive), and body weight ≥50 kg;
* Normal results of physical examination, vital signs, laboratory tests, 12 lead-ECG, chest X-ray, abdominal ultrasound, or non-clinical significance changes in the assessments above.

Exclusion Criteria:

* Subjects with a history of hypersensitivity reactions or clinically significant hypersensitivity reactions to drugs containing; or a history of allergic diseases (including but not limited to asthma, urticaria, etc.), or allergic constitution (such as known allergy to two or more substances)
* Subjects with a clear history of disorders of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic system, etc., or suggest potential diseases, such as abnormal laboratory test results of liver and kidney function (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] exceeding the upper limit of normal, or total bilirubin exceeding the upper limit of normal; Or blood creatinine exceeding the upper limit of normal value); Or other diseases (such as a history of mental illness) deemed unsuitable for participation in the trials by the investigators;
* Subjects with severe infection, severe trauma, or major surgery within 6 months prior to screening;
* Subjects who have received blood transfusions, had blood donors, or lost blood ≥400 mL within 3 months before screening; Or plan to donate blood within 1 month of the end of the trial;
* Subjects who have positive results of human immunodeficiency virus antibodies (HIV-Ab), or hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV-Ab), or syphilis specific antibodies (TPPA);
* Subjects who have participated in clinical trials for medication or medical device within 3 months prior to screening;etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (Peak Plasma Concentration (Cmax) ) of PEG-rhGH with present and new preparation | 0 hours -408 hours post-administration
Pharmacokinetics (Area under the concentration-time curve from time zero to time infinity (AUC0-inf)) of PEG-rhGH with present and new preparation | 0 hours -408 hours post-administration
Pharmacokinetics (Area under the concentration-time curve from time zero to the time of the last quantifiable (AUC0- last )) of PEG-rhGH with present and new preparation | 0 hours -408 hours post-administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China